CLINICAL TRIAL: NCT07097597
Title: Clinical Validation of a Snoring-App Compared to a Sleep Study and a Commercially Available Application
Brief Title: Validation of a Snoring App Against Commercially Available Applications and PSG
Status: Not yet recruiting | Type: Observational
Sponsor: Windsor Sleep Disorders Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ValidationSnoringApp
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Snoring; Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep Laboratory Patients
  Interventions: Device: Comparison 1: New Snoring Application; Device: Comparison 2: Commercially Available Snoring Application; Device: Comparison 3: Polysomnography

INTERVENTIONS:
Device: Comparison 1: New Snoring Application — Measurements obtained from the snoring application under development
Device: Comparison 2: Commercially Available Snoring Application — Measurements from a commercially available snoring application
Device: Comparison 3: Polysomnography — Measures taken from home or in laboratory polysomnography

SUMMARY:
This study will compare the output of a new snoring application against another commercially available application and polysomnography (either home or in-laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Referred for a diagnostic sleep study

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred for a diagnostic sleep study at the Windsor Sleep Disorders Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Snoring | 1 Night recording with all 3 devices
  Objective Measurements of snoring intensity (decibel)
Apneas | 1 Night recording with all 3 devices
  Frequency of Apneas (events per hour)
Snoring | 1 Night recording with all 3 devices
  Frequency of snoring (counts)